CLINICAL TRIAL: NCT06190899
Title: A Phase 1/2, Open-Label, Randomized, Dose Finding and Dose Expansion Study of Gedatolisib in Combination With Darolutamide in Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Brief Title: Gedatolisib in Combination With Darolutamide in Metastatic Castration-Resistant Prostate Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celcuity Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CELC-G-201
Record Dates: First submitted 2023-12-13; First posted 2024-01-05 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: mCRPC (Metastatic Castration-resistant Prostate Cancer); Genital Diseases, Male; Urogenital Diseases, Male; Prostatic Disease; Prostatic Neoplasms, Castration-Resistant; Prostate Cancer
Keywords: Gedatolisib; PI3K; Protein Kinase Inhibitors; mCRPC (metastatic castration-resistant prostate cancer); Darolutamide; Prostate Cancer; Prostatic Neoplasms, Castration-Resistant; Prostatic Disease; Urogenital Diseases, Male; Genital Diseases, Male
MeSH Terms: conditions — Genital Diseases, Male; Male Urogenital Diseases; Prostatic Diseases; Prostatic Neoplasms, Castration-Resistant; Prostatic Neoplasms | interventions — gedatolisib; darolutamide

STUDY DESIGN:
Intervention Model Description: This is a Phase 1/2, open-label, randomized, dose finding and dose expansion study to evaluate the safety, preliminary efficacy, and PK of gedatolisib in combination with darolutamide in subjects with mCRPC. The study is comprised of two phases:
  * Phase 1 Dose Finding (2 Parts)
    o Part 1: DLT evaluation and determination of tolerated doses
  * Part 2: Determination of RP2D
  * Phase 2 Dose Expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1 Arm 1 (Experimental): Arm 1 - 120 mg of gedatolisib (administered once weekly for 3 weeks on/1 week off) in combination with darolutamide 600 mg (two 300 mg tablets) orally administered twice daily (equivalent to a total daily dose of 1200 mg on Days 1-28 of each cycle)
  Interventions: Drug: Gedatolisib; Drug: Darolutamide
- Phase 1 Arm 2 (Experimental): Arm 2 - 180 mg of gedatolisib (administered once weekly for 3 weeks on/1 week off) in combination with darolutamide 600 mg (two 300 mg tablets) orally administered twice daily (equivalent to a total daily dose of 1200 mg on Days 1-28 of each cycle)
  Interventions: Drug: Gedatolisib; Drug: Darolutamide
- Phase 2 (Experimental): The recommended Phase 2 dose (RP2D) of gedatolisib (administered once weekly for 3 weeks on/1 week off) in combination with darolutamide 600 mg (two 300 mg tablets) orally administered twice daily (equivalent to a total daily dose of 1200 mg on Days 1-28 of each cycle)
  Interventions: Drug: Gedatolisib; Drug: Darolutamide

INTERVENTIONS:
Drug: Gedatolisib — Gedatolisib is a potent reversible inhibitor that selectively targets all Class I PI3K isoforms and mTOR.
Drug: Darolutamide — Darolutamide is a novel androgen receptor inhibitor that has been studied and received approval for treatment of patients with nonmetastatic CRPC and in metastatic hormone-sensitive prostate cancer.
  Other Names: NUBEQA

SUMMARY:
This is a Phase 1/2, open-label, randomized, dose finding and dose expansion study to evaluate the safety, preliminary efficacy, and PK of gedatolisib in combination with darolutamide in subjects with mCRPC.

DETAILED DESCRIPTION:
This is a Phase 1/2, open-label, randomized, dose finding and dose expansion study to evaluate the safety, preliminary efficacy, and pharmacokinetics of gedatolisib, a pan-PI3K/mTOR inhibitor, in combination with darolutamide, a next-generation androgen receptor inhibitor, in patients with metastatic castration-resistant prostate cancer following progression on a next-generation androgen receptor inhibitor. The aim of the Phase 1 portion of the study is to evaluate dose limiting toxicities and to determine the recommended Phase 2 dose. The aim of the Phase 2 portion of the study is to further assess the safety and preliminary efficacy of the drug combination.

ELIGIBILITY:
Inclusion Criteria

1. Adult males ≥18 years of age
2. Histologically or cytologically confirmed diagnosis of adenocarcinoma of the prostate without a small cell component and with <10% neuroendocrine type cells
3. Subjects must have metastatic castration-resistant prostate cancer (mCRPC; i.e., developed progression of metastases following surgical castration or during medical androgen ablation therapy)
4. Metastatic disease identified by conventional imaging: computed tomography (CT), magnetic resonance imaging (MRI), or technetium 99m-methyl diphosphonate (99mTc-MDP) bone scintigraphy. Measurable and non-measurable disease are allowed, but metastases visible only on prostate-specific membrane antigen (PSMA) positron emission tomography (PET) will not be allowed for eligibility purposes.
5. Progressive mCRPC based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 with modifications as specified in Prostate Cancer Working Group 3 (PCWG3) criteria as defined by at least one of the following criteria:

   5.1. Prostate-specific antigen (PSA) progression defined as a minimum of 2 rising PSA levels with a minimum of a 1-week interval between each determination. A minimum PSA of 1.0 ng/mL is required for study entry.

   5.2. Soft-tissue progression defined as an increase ≥20% in the sum of the longest diameter (LD) of all target lesions based on the smallest sum LD since treatment started or the appearance of one or more new lesions. 5.3. Progression of bone disease (measurable disease) or 2 or more new bone lesions by bone scan.
6. Continued primary androgen deprivation with luteinizing hormone-releasing hormone (LHRH) analog (agonist or antagonist) if the subject has not undergone bilateral orchiectomy
7. Eastern Cooperative Oncology Group (ECOG) performance status score ≤1
8. Progression during treatment with one next-generation androgen receptor signaling inhibitor for metastatic disease (e.g., abiraterone, enzalutamide, apalutamide, darolutamide)
9. Completion of prior treatment with an androgen receptor inhibitor (ARi) ≥4 weeks before the first dose of the study drug
10. At least 2 weeks beyond treatment with a targeted therapy or major surgery and at least 3 weeks beyond any other systemic anticancer therapy and/or radiation therapy, and resolution of all toxicities related to prior therapies or surgical procedures to baseline (except alopecia, Grade 1 peripheral neuropathy)
11. Adequate bone marrow, hepatic, renal and coagulation function

Exclusion Criteria

1. History of malignancies other than adequately treated non-melanoma skin cancer or other solid tumors curatively treated with no evidence of disease for ≥3 years
2. Adenocarcinoma of the prostate with a small cell component, and with ≥10% neuroendocrine type cells
3. Prior treatment with a phosphoinositide 3-kinase (PI3K) inhibitor, a protein kinase B (AKT) inhibitor, or a mechanistic target of rapamycin (mTOR) inhibitor
4. Prior treatment with chemotherapy or radiopharmaceutical therapy for mCRPC (except prior chemotherapy plus ADT for castration-sensitive disease, including docetaxel plus darolutamide).
5. Subjects with uncontrolled type 1 or type 2 diabetes

9. Known and untreated, or active, brain or leptomeningeal metastases. Subjects with previously treated central nervous system (CNS) metastases may be enrolled in the study if they meet the following criteria: do not require supportive therapy with steroids; do not have seizures and do not exhibit uncontrolled neurological symptoms; stable disease confirmed by radiographic assessment within at least 4 weeks prior to randomization 10. History of clinically significant cardiovascular abnormalities 11. Gastrointestinal tract disease resulting in an inability to absorb oral medication as well as history of inflammatory bowel disease 12. Unable to swallow oral medication tablets/capsules

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult Males
Enrollment: 54 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Assessment of the safety and tolerability of gedatolisib in combination with darolutamide in metastatic castration-resistant prostate cancer (mCRPC) | Cycle 1, Day 1 to end of safety follow up (each cycle is 28 days and safety follow up will continue until 30 days after last dose of study medication)
  Type, incidence, severity (as graded by National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] v5.0), seriousness, and relationship to study medications of adverse events (AEs) and any laboratory abnormalities
Phase 1: Identification of the recommended Phase 2 dose (RP2D) of gedatolisib in combination with darolutamide in mCRPC | Through Phase I completion, an average of 1 year.
  Incidence of dose-limiting toxicities (DLTs) and AEs graded according to NCI CTCAE v5.0
Phase 2: Assessment of the antitumor activity of gedatolisib in combination with darolutamide in each arm as demonstrated by radiographic progression-free survival (rPFS) by arm | 6 months
  Radiographic progression-free survival rate at 6 months as measured by the Kaplan-Meier (K-M) method and assessed based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 with modifications as specified in Prostate Cancer Working Group 3 (PCWG3) criteria

SECONDARY OUTCOMES:
Assessment of the preliminary efficacy of gedatolisib in combination with darolutamide by arm | 9 and 12 months post Cycle 1 Day 1 (each cycle is 28 days); 18 and 24 months post Cycle 1 Day 1 (each cycle is 28 days)
  Radiographic progression-free survival rates at 9 and 12 months and overall rPFS Overall Survival (OS) rate at 18 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Nadene Zack, MS, Study Director — Celcuity Inc
Locations (13):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States
- France (4):
  - Centre Jean Perrin, Clermont-Ferrand
  - Institut Paoli-Calmettes, Marseille
  - Centre Antoine Lacassagne, Nice
  - Institut Gustave Roussy, Villejuif
- Spain (5):
  - Hospital Clinic Barcelona, Barcelona
  - Institut Catala d'Oncologia, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital 12 de Octubre, Madrid
  - Instituto Valenciano de Oncología, Valencia
- United Kingdom (3):
  - Cambridge University Hospitals NHS Foundation Trust - Addenbrooke's Hospita, Cambridge
  - University Hospital Southampton NHS Foundation Trust - Southampton General Hospital, Southampton
  - Royal Marsden NHS Foundation Trust, Sutton